CLINICAL TRIAL: NCT06223906
Title: A Registry Study of Biomarkers in Heart Valve Disease
Acronym: BIOMS-HVD
Status: Recruiting | Type: Observational
Sponsor: Beijing Institute of Heart, Lung and Blood Vessel Diseases (Other)
Responsible Party: Sponsor
Other Study IDs: BIOMS-HVD
Record Dates: First submitted 2024-01-16; First posted 2024-01-25 (Actual); Last update posted 2024-01-26 (Actual); Status verified 2021-01

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Valvular Heart Disease, impacting 2.5% of the population, is predominantly observed in the elderly and is on the rise. The primary conditions within this category are Aortic Stenosis and Mitral Regurgitation. These conditions are linked to considerable morbidity and mortality, presenting a formidable challenge in optimizing treatment strategies. Pathophysiology of Valvular Heart Disease remains poorly known. The aim of the present study is to identify biomarkers involved in this disease using multi-omics approaches

ELIGIBILITY:
Inclusion Criteria:

* Patients clinically diagnosed with heart valve disease in Beijing Anzhen Hospital

Exclusion Criteria:

* Age < 18 years
* Failure to obtain medical records and ultrasound data
* Refuse follow-up

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with heart valve disease accorrding to Inclusion and exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 200000 (Estimated)
Dates: Start 2016-01-01 (Actual); Primary Completion 2030-01-01 (Estimated); Study Completion 2030-01-01 (Estimated)

PRIMARY OUTCOMES:
All-cause death | These data is collected during follow-up visit at 12 months after discharge
  whether recidivation happened,whether other related disease happened

SECONDARY OUTCOMES:
HF rehospitalization | These data is collected during follow-up visit at 12 months after discharge
  heart failure related hospitalization within 1 years of discharge

CONTACTS AND LOCATIONS:
Overall Officials: Jie Du, Dr, Study Director — The Key Laboratory of Remodeling-Related Cardiovascular Disease, Ministry of Education, Beijing Anzhen Hospital, Capital Medical University, Beijing Institute of Heart,Lung and Blood Vessel Diseases
Locations (1):
- Beijing Anzhen Hospital, Beijing, Beijing Municipality, China